CLINICAL TRIAL: NCT04584047
Title: Evaluation of Cell-based Non-invasive Prenatal Testing as an Alternative to Chorionic Villus Sampling as a Tool to Confirm the Pregnancy With an Unaffected Fetus Following Preimplantation Genetic Testing
Brief Title: Cell Based Non Invasive Prenatal Testing as an Alternative to Chorionic Villus Sampling Following Preimplantation Genetic Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Arcedi Biotech (Industry); Aarhus University Hospital (Other); Viborg Regional Hospital (Other); Horsens Hospital (Other); Randers Regional Hospital (Other); Kolding Sygehus (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christian Liebst Frisk Toft, Molecular Biologist, Ph.D. fellow, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N-20180001
Record Dates: First submitted 2020-09-23; First posted 2020-10-12 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Prenatal Diagnoses; Preimplantation Genetic Diagnosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): This arm has blood collected either at the time of CVS.
  Interventions: Procedure: Cell-based non-invasive prenatal testing

INTERVENTIONS:
Procedure: Cell-based non-invasive prenatal testing — Blood sampling.

SUMMARY:
The study aims to investigate whether cell-based non-invasive prenatal testing (cbNIPT) can be used as an alternative to invasive chorionic villus sampling (CVS) in patients who achieve pregnancy following preimplantation genetic testing for monogenic disorders (PGT-M).

ELIGIBILITY:
Inclusion Criteria:

* Achieved pregnancy following preimplantation genetic testing

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Agreement between cbNIPT and CVS (The gold standard) | Immidiately after the results from cbNIPT and CVS has been obtained
  How do the cbNIPT results compare to the results of the genetic test following CVS

SECONDARY OUTCOMES:
Effectiveness of fetal cell isolation | Immidiately after genetic testing of the isolated fetal cells
  How large a fraction of the potential fetal cells isolated is verified by genetic testing to be of fetal origin.
Effectiveness of testing the genetic variant of interest | Immidiately after genetic testing of the isolated fetal cells
  How often does the test on a fetal cell yield a result that allows determination of the mutational status of the embryo with respect to the genetic variant of interest.

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Unit, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD is shared upon request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon request
Access Criteria: Contact via principal investigator